CLINICAL TRIAL: NCT05948124
Title: Carnitine Deficiency and Benefits of Its Supplementation in Pediatric Hemodialysis Patients
Brief Title: Carnitine Supplementation in Pediatric Hemodialysis Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fady georguos labib, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Carnitine in Hemodialysis
Record Dates: First submitted 2023-06-17; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Carnitine Deficiency Due to Hemodialysis
MeSH Terms: interventions — Carnitine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Carnitine Group (Experimental): Enrolled patients in this group who are on regular hemodialysis fulfilling our study's inclusion criteria with secondary carnitine deficiency(based on clinical manifestations and decreased serum level of L-carnitine ;serum free carnitine level less than 20 μmol/L) will receive intravenous L-carnitine (20 mg/kg dry body weight) after each dialysis session three times weekly for 6 months.
  Interventions: Drug: L-carnitine
- Placebo Group (Placebo Comparator): enrolled patients in this group who will receive 5 ml intravenous isotonic saline after each dialysis session three times weekly for 6 months.
  Interventions: Other: isotonic saline

INTERVENTIONS:
Drug: L-carnitine — L-carnitine supplementation
  Arms: L-Carnitine Group
Other: isotonic saline — Intravenous 5 ml of isotonic saline
  Arms: Placebo Group

SUMMARY:
The goal of this study is:

1. To determine the prevalence of carnitine deficiency among pediatric patients on hemodialysis.
2. To evaluate the efficiency of carnitine supplementation in children on regular hemodialysis with carnitine deficiency in the treatment of renal anemia, cardiac dysfunction, dyslipidemia, intradialytic muscle cramps and hypotension and their quality of life.

DETAILED DESCRIPTION:
Patients on hemodialysis (HD) often have carnitine deficiency due to multiple factors; dietary intake of carnitine is decreased due to falls in appetite, total energy levels, and protein intake. In addition, accumulating evidence has linked inflammation to malnutrition, and chronic inflammation might also interrupt carnitine transfer in the intestine. Carnitine biosynthesis can also fall in patients on dialysis due to reduced biosynthesis in the kidney and limited compensation by the liver. Furthermore, because of the low molecular weight of carnitine and its high hydrophilicity and absence of protein binding, carnitine is significantly removed by the dialyzer. As in the healthy population, carnitine deficiency in patients receiving maintenance dialysis is most commonly defined as a serum free carnitine level less than 20 μmol/L .

Intravenous levocarnitine is commonly used to treat patients receiving maintenance hemodialysis who are diagnosed with carnitine deficiency since it has 100%bioavailability and does not break down into toxic metabolites. A common dose used for carnitine supplementation is 10-20 mg/kg administered after each hemodialysis session, which produces the supraphysiologic serum levels of carnitine that are required to adequately drive carnitine from the serum into skeletal muscles.

There are four principal indications for levocarnitine treatment in dialysis patients with carnitine deficiency according to the American National Kidney Foundation: (1) erythropoiesis stimulating agents resistant anemia that has not responded to the standard erythropoiesis stimulating agent dosage; (2) recurrent symptomatic hypotension during hemodialysis;(3) symptomatic cardiomyopathy or confirmed cardiomyopathy with reduced left ventricular ejection fraction and(4) fatigability and muscle weakness that undermine the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients on regular hemodialysis for more than three months with L-carnitine deficiency.
* Anemia (hemoglobin [Hb] < 11 g/dl; hematocrit [Hct] < 30%) resistant to erythropoietin defined as Anemia that require recombinant human erythropoietin (rHuEPO) doses >300 units/kg/week intravenously in spite of adequate iron stores (transferrin saturation >20%, ferritin >100 ng/mL), and without any other identifiable cause of anemia.
* Recurrent intradialytic complications (cramping, muscular pain, hypotension)
* Cardiomyopathy with reduced left ventricular ejection fraction.
* Sex: both males and females.
* Age: 16 years old or less.

Exclusion criteria:

* Patients known to be allergic to L-carnitine.
* Patients with inborn error of metabolism.
* Patients on lipid lowering therapy.
* Patients with Diabetes mellitus.
* Patients with Associated congenital heart disease.
* Patients with Thyroid disorder, or malignancy.
* Patients received L-carnitine within the past 6 months.
* Patients received Blood transfusion 4 weeks prior to study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
change in serum free carnitine level | before supplementation and after six months of supplementation.
  The investigator will measure serum free carnitine level in blood using ELISA technique.
change in cardiac functions | before supplementation and after six months of supplementation.
  The investigator will assess ejection fraction percentage by Echocardiography.
change in hemoglobin level. | before supplementation and after six months of supplementation.
  The investigator will measure hemoglobin level to assess effect of supplementation on renal anemia. and Erythropoietin dose
change in Body composition. | before supplementation and after six months of supplementation.
  using (The Fresenius Medical Care Body Composition Monitor - BCM) to assess fat composition percentiles.
change in Body composition. | before supplementation and after six months of supplementation.
  using (The Fresenius Medical Care Body Composition Monitor - BCM) to assess lean tissue index percentiles.
change in quality of life. | before supplementation and after six months of supplementation.
  assessment of quality of life using 36 -item short form survey instrument (SF- 36) questionnaire, it is a perceived quality of life assessment tool which will be used to assess general health, physical functioning, bodily pain, and mental health with a scale 0 - 100 , The lower the score the more disability.
change in Cardiac functions | before supplementation and after six months of supplementation.
  The investigator will measure fraction shortening percentage using Echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Eknoyan G, Latos DL, Lindberg J; National Kidney Foundation Carnitine Consensus Conference. Practice recommendations for the use of L-carnitine in dialysis-related carnitine disorder. National Kidney Foundation Carnitine Consensus Conference. Am J Kidney Dis. 2003 Apr;41(4):868-76. doi: 10.1016/s0272-6386(03)00110-0. PMID 12666074
- [Background] Evans A. Dialysis-related carnitine disorder and levocarnitine pharmacology. Am J Kidney Dis. 2003 Apr;41(4 Suppl 4):S13-26. doi: 10.1016/s0272-6386(03)00113-6. PMID 12751050
- [Background] KDOQI Work Group. KDOQI Clinical Practice Guideline for Nutrition in Children with CKD: 2008 update. Executive summary. Am J Kidney Dis. 2009 Mar;53(3 Suppl 2):S11-104. doi: 10.1053/j.ajkd.2008.11.017. No abstract available. PMID 19231749